CLINICAL TRIAL: NCT00840229
Title: Rotator Interval and Intra-articular Corticosteroid Injection for Adhesive Capsulitis (Frozen Shoulder): a Randomised, Double Blind, Placebo Controlled Trial
Brief Title: Rotator Interval and Intra-articular Corticosteroid Injection for Frozen Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Tore Prestegaard, MD, consultant physician, Sykehuset i Vestfold HF
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S-08546; REK (Registry Identifier: S-08546); Interne tjenester (Other); IT-avdelingen (Other: 2008/5000); Rikshospitalet HF (Other)
Record Dates: First submitted 2009-02-08; First posted 2009-02-10 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Adhesive Capsulitis
Keywords: adhesive capsulitis; corticosteroids; injection; pain
MeSH Terms: conditions — Bursitis; Pain | interventions — triamcinolone hexacetonide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 capsular & intra-articular (Experimental): corticosteroid injection (Triamcinolone) in capsule/rotator interval and intra-articular
  Interventions: Drug: Triamcinolone hexacetonide
- 2 intra-articular (Active Comparator): corticosteroid injection (Triamcinolone) intra-articular placebo injection (Lidocaine) in capsule
  Interventions: Drug: Triamcinolone hexacetonide
- 3 placebo (Placebo Comparator): placebo injections (Lidocaine) in capsule and intra-articular
  Interventions: Drug: Triamcinolone hexacetonide

INTERVENTIONS:
Drug: Triamcinolone hexacetonide — 20 mg
  Arms: 3 placebo
Drug: Triamcinolone hexacetonide — 1 ml (20 mg) + 6 ml Lidocaine 10 mg/ml
  Arms: 1 capsular & intra-articular; 2 intra-articular

SUMMARY:
The purpose of this study is to compare ultrasound guided capsular corticosteroid injection into the rotator interval/anterior capsule and the GH joint with ultrasound guided corticosteroid injection into the GH joint only. Both methods will be compared with placebo injections.

Primary outcome measure: pain reduction at week 6 Secondary outcome measures: improvement of function (SPADI, Life quality, ROM).

0-hypothesis: no difference between the methods.

The investigators want to find out if the clinical effect of the combined capsular and intra-articular injections are better than placebo and better that intra-articular injections

DETAILED DESCRIPTION:
3 groups, 50 patients in each, follow-up visits after 3, 6, 12 and 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pain and stiffness in one shoulder 1 - 6 months
* Restriction of passive ROM; >= 30 degrees in two or more planes compared to other shoulder

Exclusion Criteria:

* Systemic inflammatory disease
* Corticosteroid treatment last 3 months
* Poorly controlled Diabetes mellitus
* Pregnancy
* Contraindications/allergy to corticosteroids and/or Lidocaine
* Severe infections
* Osteoarthritis of the shoulder
* Fractures of the shoulder
* Rotator cuff pathology causing pain or disability
* Fibromyalgia
* Not able to understand Norwegian

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2009-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Pain reduction | 2-3 years

SECONDARY OUTCOMES:
Function (ROM, SPADI), Life quality | 2-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tore A Prestgaard, MD, Principal Investigator — The Hospital of Vestfold
Locations (1):
- Vestfold Hospitalt Trust, Clinic Physical Medicine and Rehabilitation, Stavern, Norway

REFERENCES:
- [Derived] Prestgaard T, Wormgoor MEA, Haugen S, Harstad H, Mowinckel P, Brox JI. Ultrasound-guided intra-articular and rotator interval corticosteroid injections in adhesive capsulitis of the shoulder: a double-blind, sham-controlled randomized study. Pain. 2015 Sep;156(9):1683-1691. doi: 10.1097/j.pain.0000000000000209. PMID 25919473